CLINICAL TRIAL: NCT00680888
Title: Adherence in Adolescents and Children Treated on Quetiapine
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: JAVIER JIMENEZ / MEDICAL DIRECTOR, AstraZeneca Pharmaceuticals Spain S.A
Other Study IDs: NIS-NES-SER-2006/1
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Psychosis
Keywords: Psychosis; adolescents; adherence; quetiapine
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children and adolescents with psychosis in outpatients setting on treatment with quetiapine started from january 2003 to june 2006

SUMMARY:
Observational study aimed to describe the adherence in a population of adolescents and children treated on quetiapine from a first psychotic episode whose more important secondary objective is to identify possible predictive factors influencing the adherence to treatment with Quetiapine

ELIGIBILITY:
Inclusion Criteria:

* At least one psychotic symptom (delusions or hallucinations) before age 18.
* Start of treatment in a maximum period of 2 years after the onset of first psychotic symptom
* Written informed consent by parents or guardians and patients.

Exclusion Criteria:

* Pregnancy or lactancy
* High risk of aggression or suicidal behaviour
* Alcohol dependence

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents with psychosis in outpatients setting on treatment with quetiapine started from january 2003 to june 2006
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Survival analysis of rate of adherence to treatment on quetiapine | 6 months

SECONDARY OUTCOMES:
Survival analysis of rate of adherence to treatment on quetiapine | 12 months
Clinical and sociodemographic parameters (CGI-C, CGI-Suicidal, PANSS, HDRS, YMRS, SDQ, DAS, GAF, SUMD) possibly influencing adherence | 0, 6, 12 months
Tolerability profile (UKU) possibly influencing adherence | 0, 6, 12 months